CLINICAL TRIAL: NCT01893450
Title: Comparison of the Effect of Bromocriptine and Pentoxifylline in Mild to Moderate Autoimmune Ophthalmopathy. A Randomized, Controlled, Single Blind, Clinical Trial.
Brief Title: Bromocriptine and Pentoxifylline in Ophthalmopathy Autoimmune Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Efficacy demonstrated on a preliminary analysis
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Paloma Almeda-Valdés, MD, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DIA19508091
Record Dates: First submitted 2013-06-28; First posted 2013-07-09 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-07

CONDITIONS: Graves Ophthalmopathy
Keywords: Graves ophthalmopathy; Exophthalmos; Proptosis; Quality of life
MeSH Terms: conditions — Graves Ophthalmopathy; Exophthalmos | interventions — Methimazole; Bromocriptine; Pentoxifylline

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- methimazole (Active Comparator): methimazole 30 mg daily during one year
  Interventions: Drug: Methimazole
- methimazole, bromocriptine (Active Comparator): methimazole 30 mg daily during one year, bromocriptine 5 mg twice a day during one year
  Interventions: Drug: Bromocriptine
- pentoxifylline (Active Comparator): methimazol 30 mg daily and pentoxifylline 400 mg twice a day during one year
  Interventions: Drug: Pentoxifylline

INTERVENTIONS:
Drug: Methimazole
  Arms: methimazole
Drug: Bromocriptine
  Arms: methimazole, bromocriptine
Drug: Pentoxifylline
  Arms: pentoxifylline

SUMMARY:
Autoimmune ophthalmopathy is clinically evident in one third of Graves' disease cases. In most cases it is mild; however, in 3 to 5% of cases it has a severe presentation. At present, the treatment is directed to identify vision threatening which requires aggressive intervention, usually with glucocorticoids. For mild cases the treatment is limited to the normalization of hyperthyroidism and support measures. Preliminary data show that pentoxifylline and bromocriptine may have a favorable effect in the course of ophthalmopathy by inhibition of the synthesis of TNF-α, VEGF, glycosaminoglycan production, and lymphocyte infiltration. Therefore, the aims of this study were to evaluate the effect of bromocriptine and pentoxifylline on the clinical course and quality of life of patients with mild to moderate ophthalmopathy associated to Graves´disease.

Methods. Patients with mild to moderate ophthalmopathy, with less than one year of evolution, and naive to treatment were randomized to receive treatment during 12 months with either 1) bromocriptine (5 mg twice a day) + methimazole (30 mg/day), 2) pentoxifylline (400 mg twice a day) + methimazole (30 mg/day), or 3) methimazole only (30 mg/day). They completed 10 visits to evaluate proptosis and clinical activity score (CAS). In addition, in the first and last visit the quality of life questionnaire specific for Graves' ophthalmopathy(GO-QOL) was applied.

ELIGIBILITY:
Inclusion Criteria:

* Women or men
* Between 18 and 45 years
* Autoimmune hyperthyroidism with one year or less of evolution
* No previous treatment
* Mild to moderate ophthalmopathy

Exclusion Criteria:

* Smoking
* Severe ophthalmopathy
* Steroid treatment
* Asthma
* Diabetes or other significant disease
* Creatine >1.5 mg/dl
* Women with child bearing potential not using a birth control method
* Opthalmologic diseases
* Uncontrolled hypertension
* History of ischemic cardiopathy
* History of stroke
* History of gastrointestinal bleeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2008-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Proptosis | One year
  Left and right eye proptosis by exophthalmometry

SECONDARY OUTCOMES:
Clinical activity score | One year
  Clinical activity score for Graves' ophthalmopathy
Quality of life | One year
  Quality of life assessed with the quality of life questionnaire specific for Graves' ophthalmopathy (GO-QOL)

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico City, Mexico